CLINICAL TRIAL: NCT01762800
Title: Evaluating the Control of COPD Symptoms in Patients Treated With Tiotropium Bromide 18mcg Once Daily Alone, ADOAIR 50/250mcg Twice Daily Alone or ADOAIR 50/250mcg Plus Tiotropium Bromide 18mcg
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 116717
Record Dates: First submitted 2012-12-06; First posted 2013-01-08 (Estimated); Results first posted 2016-11-10 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone; Salmeterol Xinafoate; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- fluticasone propionate/salmeterol (Experimental): Randomised treatment at Visit 2
  Interventions: Drug: fluticasone propionate/salmeterol 50/250mcg; Drug: tiotropium bromide placebo; Drug: fluticasone propionate/salmeterol 50/250mcg and tiotropium 18mcg
- tiotropium bromide (Experimental): Randomised treatment at Visit 2
  Interventions: Drug: fluticasone propionate/salmeterol placebo; Drug: tiotropium bromide 18mcg; Drug: fluticasone propionate/salmeterol 50/250mcg and tiotropium 18mcg

INTERVENTIONS:
Drug: fluticasone propionate/salmeterol 50/250mcg — Active, 50/250mcg, Twice daily (morning and evening)
  Other Names: ADOAIR is a registered trade mark of the GlaxoSmithKline group of companies
  Arms: fluticasone propionate/salmeterol
Drug: fluticasone propionate/salmeterol placebo — Placebo, Twice daily (morning and evening)
  Arms: tiotropium bromide
Drug: tiotropium bromide 18mcg — Active, 18mcg, Once daily(morning)
  Arms: tiotropium bromide
Drug: tiotropium bromide placebo — Placebo, Once daily(morning)
  Arms: fluticasone propionate/salmeterol
Drug: fluticasone propionate/salmeterol 50/250mcg and tiotropium 18mcg — Active. The randomized treatment may be switched to TRIPLE therapy when COPD symptoms are uncontrolled or the subject is not satisfied with the randomized treatment at each scheduled or unscheduled visit.
  Other Names: TRIPLE therapy

SUMMARY:
The purpose of this study is to assess the control of COPD using a symptom and exacerbation risk based treatment strategy based on GOLD 2011. This study is conducted in Japanese subjects with COPD and assess whether the GOLD 2011 strategy is effective in medical practice in Japan.

DETAILED DESCRIPTION:
PROTOCOL SUMMARY Rationale Both ADOAIR and tiotropium bromide ( hereinafter tiotropium）are now well established, effective treatments for COPD and are frequently co-prescribed (hereinafter TRIPLE therapy). The addition of ADOAIR to tiotropium improves lung function and quality of life and may further reduce exacerbations. GOLD 2011 thus recommends TRIPLE therapy as the second choice of COPD treatment strategy. However, the criteria for switching from each individual treatment to TRIPLE therapy are not clearly shown so far.

This study will be conducted in Japanese subjects with COPD and will assess whether the GOLD 2011 strategy is effective in medical practice in Japan.

Objective(s) The objective of the study is to assess the control of COPD using a symptom and exacerbation risk based treatment strategy based on GOLD 2011.

Study Design Multicenter, randomized, double-dummy, 24-weeks, observational study Study Endpoints/Assessments Primary

* Proportion of patients who were able to remain on the randomized therapy Secondary
* Proportion of patients who switched to TRIPLE therapy
* Proportion of patients who controlled by TRIPLE therapy
* Proportion of patients controlled by randomized therapy plus TRIPLE therapy
* Time to switching to TRIPLE therapy
* Time to first exacerbation
* Proportion of diagnosed exacerbation confirmed by Daily Record Card
* Proportion of exacerbations detected by Daily Record Card not diagnosed
* CAT score change
* Change in FEV1
* Use of relief medication
* Proportion of patients who decreased treatment from TRIPLE therapy
* Proportion of patients who required additional treatment to TRIPLE therapy
* Proportion of patients who dropped out
* Patients' judgment of treatment efficacy
* Physician's judgment of treatment efficacy

Safety

* Adverse event reporting
* Exacerbations of COPD

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 40 - 80 years inclusive
2. Has an established clinical history of COPD (defined as per the GOLD definition)
3. The subject achieves a grade of ≥1 on mMRC at Visit 1
4. A signed and dated written informed consent is obtained from the subject prior to study participation
5. The subject has a post-bronchodilator FEV1 of ≥ 30% to ≤ 80% of predicted normal
6. The subject has a post-bronchodilator FEV1 / FVC ratio < 70%
7. The subject is a current or ex-smoker with a smoking history of > 10 pack-years Ex-smokers are required to have stopped smoking for at least 6 months prior to visit 1. Ex-smokers who stopped smoking less than 6 months ago will be defined as current smokers.
8. QTc < 450 msec at Visit 1; or for patients with bundle branch block QTc should be < 480 msec.

(QTc(F) < 450 msec, or < 480 msec in subjects with right bundle branch block, should be confirmed by the mean of three readings or one reading) 9. ALT < 2 x ULN and bilirubin/ALP ≤ 1.5 x ULN (> 35% direct bilirubin) 10. A female is eligible to enter this study if she is: i) of non-childbearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is post-menopausal), or ii) of child-bearing potential, but has a negative urinary pregnancy test at screening and agrees to take contraceptive precautions (including abstinence) which are adequate to prevent pregnancy during the study iii) not a nursing mother

Exclusion Criteria:

1. Has a predominant asthma (comorbid asthma is not an exclusion criteria)
2. Has a medical diagnosis of narrow-angle glaucoma, prostatic hyperplasia or bladder neck obstruction that in the opinion of the investigator should prevent them from entering the study Note: As with other anticholinergic drugs, subjects with narrow-angle glaucoma, prostatic hyperplasia or bladder neck obstruction should only be entered into the study at the Investigator's discretion
3. Has known respiratory disorders other than COPD (e.g. lung cancer, sarcoidosis, tuberculosis or lung fibrosis)
4. Has undergone lung surgery e.g., lung transplant and/or lung volume reduction
5. Had a chest X-ray indicating diagnosis other than COPD that might interfere with the study (chest X-ray to be taken at Visit 1, if subject has not had one and/or CT image taken within 3 months of Visit 1)
6. Requires regular (daily) or long term oxygen therapy (LTOT). (LTOT is defined as ≥ 12 hours oxygen use per day)
7. Has plan to start or to change the pulmonary rehabilitation program during the study period
8. Requires regular treatment with oral, parenteral, or depot corticosteroids
9. Has serious, uncontrolled disease likely to interfere with the study (e.g. Left Ventricular failure, anaemia, renal or hepatic disease or serious psychological disorders)
10. Received any other investigational drugs within 4 weeks (or 5 half lives) prior to Visit 1
11. Has, in the opinion of the investigator, evidence of alcohol, drug or solvent abuse
12. Has a known or suspected hypersensitivity to β2-agonists, steroids, anticholinergic treatments or any components of the formulations
13. Has previously been enrolled to this study and investigational drugs has been administered
14. Is not eligible to participate this study in the opinion of the investigator/subinvestigator

The investigator must refer to the following document(s) for detailed information regarding warnings, precautions, contraindications, adverse events, and other significant data pertaining to the investigational product(s) being used in this study:

1. ADOAIR DISKUS package insert
2. Tiotropium/ HandiHaler package insert
3. Salbutamol package insert

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2013-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (17):
- Japan (17):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kochi
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Nara
  - GSK Investigational Site, Niigata
  - GSK Investigational Site, Okinawa
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Saga
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Yamaguchi

REFERENCES:
- [Derived] Betsuyaku T, Kato M, Fujimoto K, Hagan G, Kobayashi A, Hitosugi H, James M, Jones PW. A study to assess COPD Symptom-based Management and to Optimise treatment Strategy in Japan (COSMOS-J) based on GOLD 2011. Int J Chron Obstruct Pulmon Dis. 2013;8:453-9. doi: 10.2147/COPD.S48298. Epub 2013 Oct 3. PMID 24124358

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 570 participants were screened, 428 participants entered into the run-in period, 406 participants were randomized into the study (incorrectly 407 on protocol summary due to miss operation at study site that cannot be corrected), and 405 participant received study medication and comprised the modified Intent to Treat (mITT) Population.
Groups:
- TIO 18 µg QD: Participants received 18 micrograms (µg) tiotropium bromide (TIO) once daily (QD) via HandiHaler inhaler and placebo twice daily (BID) via dry powder inhaler (DPI), during the 24-week study treatment period. Participants also received 400 µg salbutamol as relief medication and as a bronchodilator for pulmonary function testing as required throughout the study.
- SAL/FLU 50/250 µg BID: Participants received 50/250 µg salmeterol xinafoate (SAL)/fluticasone propionate (FLU) BID via DPI and placebo QD via HandiHaler inhaler, during the 24-week study treatment period. Participants also received 400 µg salbutamol as relief medication and as a bronchodilator for pulmonary function testing as required throughout the study.
Period: Overall Study
Arm/Group | TIO 18 µg QD | SAL/FLU 50/250 µg BID
Started | 202 | 204
Completed | 183 | 183
Not Completed | 19 | 21
Not completed — Adverse Event | 8 | 13
Not completed — Lack of Efficacy | 3 | 2
Not completed — Study Closed/Terminated | 0 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 7 | 4

BASELINE CHARACTERISTICS:
Population: 406 participants were randomized into the study, however 405 participant received study mediciation and comprised the modified Intent to Treat (mITT) Population.
Groups:
- TIO 18 µg QD: Participants received 18 µg TIO QD via HandiHaler inhaler and placebo BID via DPI, during the 24-week study treatment period. Participants also received 400 µg salbutamol as relief medication and as a bronchodilator for pulmonary function testing as required throughout the study.
- SAL/FLU 50/250 µg BID: Participants received 50/250 µg SAL/FLU BID via DPI and placebo QD via HandiHaler inhaler, during the 24-week study treatment period. Participants also received 400 µg salbutamol as relief medication and as a bronchodilator for pulmonary function testing as required throughout the study.
- Total: Total of all reporting groups
Arm/Group | TIO 18 µg QD | SAL/FLU 50/250 µg BID | Total
Number analyzed (Participants) | 201 | 204 | 405
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.0 (7.12) | 68.6 (6.93) | 68.3 (7.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 20
  Male | 193 | 192 | 385
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 0 | 1 | 1
  Asian - Japanese Heritage | 201 | 203 | 404

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Were Able to Remain on the Randomized Treatment
Description: The randomized treatment could be switched to TRIPLE therapy in the case that chronic obstructive pulmonary disease (COPD) is not controlled by the randomized treatment. Participants on TRIPLE therapy received SAL/FLU 50/250 µg BID plus TIO 18 µg QD together. The percentage of participants who were able to remain on the randomized treatment was calculated by the following formula: 100 minus percentage of participants who switched over to TRIPLE therapy.
Time Frame: 24 weeks
Population: Modified Intent-to-Treat (mITT) population: randomized participants who received at least a single dose of the investigational product.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TIO 18 µg QD | SAL/FLU 50/250 µg BID
Number analyzed (Participants) | 201 | 204
Percentage of participants | 62.69 [55.60 to 69.39] | 66.67 [59.75 to 73.10]

2. Secondary Outcome: Percentage of Participants Who Switched to TRIPLE Therapy
Description: Switched to TRIPLE therapy is defined as: 1. Date of switch: when SAL/FLU or TIO was administered additionally to randomised treatment. 2. Date of randomisation was a start point and timing of switching (first switch if there are more than once) to TRIPLE was event. For participants without switching, last day of study or follow up period was regarded as censored. Percentage of participants who switched to TRIPLE therapy was calculated as: number of participants who switched to TRIPLE therapy divided by number of evaluable population and then multiplied by 100.
Time Frame: 24 weeks
Population: mITT population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TIO 18 µg QD | SAL/FLU 50/250 µg BID
Number analyzed (Participants) | 201 | 204
Percentage of participants | 37.31 [30.61 to 44.40] | 33.33 [26.90 to 40.25]

3. Secondary Outcome: Percentage of Participants Managed by TRIPLE Therapy
Description: Percentage of participants managed by TRIPLE therapy was calculated as [(number of participants who switched to TRIPLE therapy) - (number of participants who stepped down)/ number of evaluable population]*100
Time Frame: 24 weeks
Population: mITT population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TIO 18 µg QD | SAL/FLU 50/250 µg BID
Number analyzed (Participants) | 201 | 204
Percentage of participants | 36.82 [30.14 to 43.89] | 32.35 [25.99 to 39.24]

4. Secondary Outcome: Continuation Percentage of Participants Managed by Randomized Treatment Plus TRIPLE Therapy
Description: The randomized treatment could be switched to TRIPLE therapy in the case that chronic obstructive pulmonary disease (COPD) was not controlled by the randomized treatment. Participants on TRIPLE therapy received SAL/FLU 50/250 µg BID plus TIO 18 µg QD together. Continuation TRIPLE proportion is defined as [(number of subjects who switched to TRIPLE) - (number of subjects who stepped down)/ number of evaluable population]*100. Randomised treatment continuation proportion is calculated by a formula: (100 - switch proportion).
Time Frame: 24 weeks
Population: mITT population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TIO 18 µg QD | SAL/FLU 50/250 µg BID
Number analyzed (Participants) | 201 | 204
Percentage of participants
  Randomised treatment | 62.69 [55.60 to 69.39] | 66.67 [59.75 to 73.10]
  TRIPLE therapy | 36.82 [30.14 to 43.89] | 32.35 [25.99 to 39.24]

5. Secondary Outcome: Time to First Switching to TRIPLE Therapy
Description: The day of first switch to TRIPLE therapy (SAL/FLU 50/250 µg BID+TIO 18 µg QD) for the first switching participant in each arm.
Time Frame: 24 weeks
Population: mITT population
Measure: Number; unit: Days
Arm/Group | TIO 18 µg QD | SAL/FLU 50/250 µg BID
Number analyzed (Participants) | 201 | 204
Days | 5 | 5

6. Secondary Outcome: Time to First Exacerbation by Physician's Diagnosis
Description: The day of detection of first exacerbation in any participant in each arm as diagnosed by physician. Exacerbation is defined primarily by physician's judgment. Date of randomisation will be start point and timing of exacerbation (first exacerbation if there are more than one) will be event. For subjects without exacerbation, last day of study or follow up period is regarded as censor.
Time Frame: 24 weeks
Population: mITT population
Measure: Number; unit: Days
Groups:
- SAL/FLU 50/250 µg BID-Single: Participants received 50/250 µg SAL/FLU BID via DPI and placebo QD via HandiHaler inhaler, during the 24-week study treatment period. Participants also received 400 µg salbutamol as relief medication and as a bronchodilator for pulmonary function testing as required throughout the study. Participants who remained on the single treatment of SAL/FLU 50/250 µg BID were included in this arm.
- SAL/FLU 50/250 µg BID-TRIPLE: Participants received 50/250 µg SAL/FLU BID via DPI and placebo QD via HandiHaler inhaler, during the 24-week study treatment period. Participants also received 400 µg salbutamol as relief medication and as a bronchodilator for pulmonary function testing as required throughout the study. Participants who switched from the single treatment of SAL/FLU 50/250 µg BID to TRIPLE therapy (SAL/FLU 50/250 µg BID+TIO 18 µg QD) were included in this arm.
- TIO 18 µg QD-Single: Participants received 18 µg TIO QD via HandiHaler inhaler and placebo BID via DPI, during the 24-week study treatment period. Participants also received 400 µg salbutamol as relief medication and as a bronchodilator for pulmonary function testing as required throughout the study. Participants who remained on the single treatment of TIO 18 µg QD were included in this arm.
- TIO 18 µg QD-TRIPLE: Participants received 18 µg TIO QD via HandiHaler inhaler and placebo BID via DPI, during the 24-week study treatment period. Participants also received 400 µg salbutamol as relief medication and as a bronchodilator for pulmonary function testing as required throughout the study. Participants who switched from the single treatment of TIO 18 µg QD to TRIPLE therapy (SAL/FLU 50/250 µg BID+TIO 18 µg QD) were included in this arm.
Arm/Group | SAL/FLU 50/250 µg BID-Single | SAL/FLU 50/250 µg BID-TRIPLE | TIO 18 µg QD-Single | TIO 18 µg QD-TRIPLE
Number analyzed (Participants) | 136 | 68 | 126 | 75
Days | 3 | 5 | 10 | 2

7. Secondary Outcome: Time to First Exacerbation by EXAcerbations of Chronic Pulmonary Disease Tool (EXACT)
Description: The EXAcerbations of Chronic pulmonary disease Tool (EXACT) is a 14-item patient-reported outcome (PRO) daily diary used to quantify and measure exacerbations of chronic obstructive pulmonary disease (COPD). Reported as units on a 0 [best health status] to 100 [worst possible status] scale). The day of detection of first exacerbation in any participant in each arm by EXACT.
Time Frame: 24 weeks
Measure: Number; unit: Days
Arm/Group | SAL/FLU 50/250 µg BID-Single | SAL/FLU 50/250 µg BID-TRIPLE | TIO 18 µg QD-Single | TIO 18 µg QD-TRIPLE
Number analyzed (Participants) | 136 | 68 | 126 | 75
Days | 0 | 0 | 0 | 1

8. Secondary Outcome: EXACT Total Score.
Description: EXACT is a 14-item patient questionnaire used as a measure of respiratory symptoms (reported as units on a 0 [best health status] to 100 [worst possible status] scale). Scores were assessed at Baseline, Week 1-4, Week 5-8, Week 9-12, Week 13-16, Week 17-20 and Week 21-24. Daily EXACT total score is obtained as total score of 14 items from diary. Daily E-RS total score as 11 items and Daily E-RS subscale scores are subset of E-RS total score.
  Mean EXACT total score is mean value of daily EXACT total score within subject by every 4 weeks(Week1-4, Week5-8, Week9-12, Week13-16, Week17-20, Week21-24). Same calculation of mean values are applied to E-RS total and E-RS subscale scores.
Time Frame: Baseline and up to 24 weeks
Population: mITT population. Only those participants available at the specified time points (represented by n=X, X, X, X in the category titles) were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SAL/FLU 50/250 µg BID-Single | SAL/FLU 50/250 µg BID-TRIPLE | TIO 18 µg QD-Single | TIO 18 µg QD-TRIPLE
Number analyzed (Participants) | 136 | 68 | 126 | 75
Scores on a scale
  Baseline; n=125, 66, 111, 71 | 28.99 (10.151) | 36.00 (10.499) | 29.77 (10.163) | 35.78 (9.222)
  Week 1-4; n=120, 67, 109, 73 | 27.83 (10.225) | 36.92 (10.385) | 28.88 (10.182) | 38.26 (12.230)
  Week 5-8; n=117, 63, 102, 69 | 27.35 (10.921) | 37.58 (9.831) | 28.80 (10.274) | 35.87 (11.117)
  Week 9-12; n=109, 67, 101, 72 | 27.63 (11.847) | 36.16 (11.492) | 28.40 (9.619) | 35.57 (11.578)
  Week 13-16; n=105, 65, 100, 71 | 27.33 (10.715) | 35.92 (11.550) | 28.93 (9.721) | 33.79 (12.334)
  Week 17-20; n=107, 65, 97, 66 | 26.98 (10.971) | 34.92 (10.661) | 28.66 (10.970) | 34.03 (12.066)
  Week 21-24; n=79, 51, 77, 46 | 26.50 (11.697) | 32.72 (11.992) | 28.80 (10.497) | 33.67 (12.722)

9. Secondary Outcome: EXACT Respiratory Symptoms (E-RS) Total Score
Description: The E-RS total score is an 11-item patient questionnaire, which provides information specific to respiratory symptoms-severity of respiratory symptoms overall and severity of breathlessness, cough and sputum, and chest symptoms. Scores were assessed at Baseline, Week 1-4, Week 5-8, Week 9-12, Week 13-16, Week 17-20 and at Week 21-24. Daily EXACT total score is obtained as total score of 14 items from diary. Daily E-RS total score as 11 items and Daily E-RS subscale scores are subset of E-RS total score.
  Mean EXACT total score is mean value of daily EXACT total score within subject by every 4 weeks(Week1-4, Week5-8, Week9-12, Week13-16, Week17-20, Week21-24). Same calculation of mean values are applied to E-RS total and E-RS subscale scores. Scores range from 0-100, high value in score indicate worse outcome.
Time Frame: Baseline and up to 24 weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SAL/FLU 50/250 µg BID-Single | SAL/FLU 50/250 µg BID-TRIPLE | TIO 18 µg QD-Single | TIO 18 µg QD-TRIPLE
Number analyzed (Participants) | 136 | 68 | 126 | 75
Scores on a scale
  Baseline; n=135, 67, 124, 73 | 7.42 (5.541) | 11.43 (6.378) | 7.51 (5.583) | 11.36 (5.650)
  Week 1-4; n=131, 68, 121, 75 | 6.76 (5.405) | 12.39 (6.533) | 7.18 (5.745) | 13.23 (7.370)
  Week 5-8; n=126, 68, 115, 73 | 6.75 (5.618) | 11.86 (6.573) | 6.99 (5.720) | 11.11 (6.798)
  Week 9-12; n=122, 68, 116, 74 | 6.69 (6.489) | 11.79 (6.696) | 6.70 (5.244) | 11.30 (6.762)
  Week 13-16; n=121, 66, 116, 74 | 6.23 (5.667) | 11.66 (6.739) | 6.82 (5.392) | 10.26 (7.122)
  Week 17-20; n=118, 66, 114, 72 | 6.33 (5.786) | 10.80 (6.158) | 6.85 (6.035) | 9.89 (7.073)
  Week 21-24; n=93, 51, 94, 51 | 5.99 (6.044) | 9.82 (6.507) | 6.58 (5.702) | 9.59 (7.420)

10. Secondary Outcome: E-RS Subscale Score
Description: The E-RS total score is an 11-item patient questionnaire, which provides information specific to respiratory symptoms-severity of respiratory symptoms overall and severity of breathlessness, cough and sputum, and chest symptoms. The E-RS subscale scores for respiratory symptoms (RS)-breathlessness (RS-BRL), RS-cough and sputum (RS-CSP), and RS-chest symptoms (RS-CSY) are presented. Scores were assessed at Baseline, Week 1-4, Week 5-8, Week 9-12, Week 13-16, Week 17-20 and at Week 21-24. Daily EXACT total score is obtained as total score of 14 items from diary. Daily E-RS total score as 11 items and Daily E-RS subscale scores are subset of E-RS total score. Mean EXACT total score is mean value of daily EXACT total score within subject by every 4 weeks(Week1-4, Week5-8, Week9-12, Week13-16, Week17-20, Week21-24). Same calculation of mean values are applied to E-RS total and E-RS subscale scores. RS total scores range from 0 to 40, high value in score indicate worse outcome.
Time Frame: 24 weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SAL/FLU 50/250 µg BID-Single | SAL/FLU 50/250 µg BID-TRIPLE | TIO 18 µg QD-Single | TIO 18 µg QD-TRIPLE
Number analyzed (Participants) | 136 | 68 | 126 | 75
Scores on a scale
  RS-BRL; Baseline; n=135, 68, 125, 73 | 3.36 (3.113) | 5.81 (3.542) | 3.41 (3.122) | 5.62 (3.393)
  RS-BRL; Week 1-4; n=131, 68, 121, 75 | 3.06 (3.245) | 6.28 (3.498) | 3.36 (3.288) | 6.59 (4.191)
  RS-BRL; Week 5-8; n=126, 68, 115, 73 | 3.08 (3.281) | 5.96 (3.517) | 3.18 (3.110) | 5.38 (3.857)
  RS-BRL; Week 9-12; n=122, 68, 116, 74 | 3.08 (3.402) | 5.87 (3.612) | 2.98 (2.970) | 5.52 (3.793)
  RS-BRL; Week 13-16; n=121, 66, 116, 74 | 2.80 (3.151) | 5.81 (3.683) | 3.04 (3.084) | 5.11 (4.029)
  RS-BRL; Week 17-20; n=118, 66, 114, 72 | 2.82 (3.349) | 5.56 (3.678) | 3.04 (3.254) | 4.94 (3.908)
  RS-BRL; Week 21-24; n=93, 51, 94, 51 | 2.79 (3.316) | 4.94 (3.661) | 2.95 (3.160) | 4.71 (4.159)
  RS-CSP; Baseline; n=135, 68, 124, 73 | 2.29 (1.536) | 2.73 (1.778) | 2.23 (1.643) | 2.81 (1.601)
  RS-CSP; Week 1-4; n=131, 68, 121, 75 | 2.12 (1.453) | 2.90 (1.687) | 2.13 (1.517) | 3.05 (1.925)
  RS-CSP; Week 5-8; n=126, 68, 116, 73 | 2.03 (1.448) | 2.83 (1.814) | 2.13 (1.633) | 2.74 (1.763)
  RS-CSP; Week 9-12; n=122, 68, 116, 74 | 2.06 (1.850) | 2.81 (1.766) | 2.11 (1.635) | 2.77 (1.803)
  RS-CSP; Week 13-16; n=121, 66, 116, 74 | 1.98 (1.563) | 2.74 (1.769) | 2.09 (1.579) | 2.49 (1.797)
  RS-CSP; Week 17-20; n=119, 66, 114, 72 | 2.06 (1.612) | 2.43 (1.608) | 2.09 (1.702) | 2.40 (1.768)
  RS-CSP; Week 21-24; n=93, 51, 94, 51 | 1.82 (1.711) | 2.27 (1.604) | 1.99 (1.680) | 2.34 (1.783)
  RS-CSY; Baseline; n=135, 67, 125, 73 | 1.77 (1.768) | 2.93 (1.903) | 1.84 (1.729) | 2.92 (1.794)
  RS-CSY; Week 1-4; n=131, 68, 121, 75 | 1.58 (1.652) | 3.21 (2.071) | 1.69 (1.681) | 3.59 (2.306)
  RS-CSY; Week 5-8; n=126, 68, 116, 73 | 1.65 (1.760) | 3.05 (1.977) | 1.70 (1.695) | 2.99 (2.149)
  RS-CSY; Week 9-12; n=122, 68, 116, 74 | 1.54 (2.032) | 3.12 (2.069) | 1.60 (1.584) | 3.01 (2.204)
  RS-CSY; Week 13-16; n=121, 66, 116, 74 | 1.46 (1.752) | 3.11 (2.102) | 1.70 (1.623) | 2.66 (2.184)
  RS-CSY; Week 17-20; n=119, 66, 114, 72 | 1.48 (1.802) | 2.81 (1.873) | 1.72 (1.908) | 2.55 (2.171)
  RS-CSY; Week 21-24; n=93, 51, 94, 51 | 1.38 (1.944) | 2.61 (1.988) | 1.64 (1.741) | 2.53 (2.167)

11. Secondary Outcome: Comparison of Number of Exacerbations Between Two Detection Methods: EXACT and Physician Diagnosis
Description: The comparison of number of exacerbation between two detection methods EXACT and physician diagnosis: number of exacerbations detected by EXACT and number of exacerbations judged by physician.
Time Frame: 24 weeks
Population: mITT population
Measure: Mean (Standard Deviation); unit: Number of exacerbations
Arm/Group | TIO 18 µg QD | SAL/FLU 50/250 µg BID
Number analyzed (Participants) | 201 | 204
Number of exacerbations
  EXACT | 0.9 (1.00) | 0.7 (1.06)
  Physician's diagnosis | 0.2 (0.44) | 0.1 (0.36)

12. Secondary Outcome: Chronic Obstructive Pulmonary Disease (COPD) Assessment Test (CAT) Total Score
Description: Participants were assessed for COPD symptoms by means of CAT at each Visit. This assessment was performed prior to the spirometry testing. A CAT total score of less than 10 represents best health status and greater than 15 represents worst health status. Scores were assessed at Visit 1 (Screening), Visit 2 (Baseline), Visit 3 (Week 4), Visit 4 (Week 8), Visit 5 (Week 8), Visit 6 (Week 12), Visit 7 (Week 16), and Visit 8 (Week 24). Scores range from 0 to 40, high value in score indicate worse outcome.
Time Frame: 24 weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SAL/FLU 50/250 µg BID-Single | SAL/FLU 50/250 µg BID-TRIPLE | TIO 18 µg QD-Single | TIO 18 µg QD-TRIPLE
Number analyzed (Participants) | 136 | 68 | 126 | 75
Scores on a scale
  Visit 1, n=136, 68, 126, 75 | 11.3 (5.83) [lower limit 5.83] | 13.3 (6.35) | 11.2 (5.77) | 13.4 (6.49)
  Visit 2, n=136, 68, 126, 75 | 9.9 (6.35) [lower limit 6.35] | 13.4 (7.52) | 9.6 (6.27) | 12.1 (6.08)
  Visit 3, n=132, 68, 121, 75 | 8.4 (6.09) [lower limit 6.09] | 13.5 (8.12) | 9.2 (5.91) | 14.3 (7.28)
  Visit 4, n=127, 68, 116, 74 | 8.3 (5.99) [lower limit 5.99] | 13.2 (7.59) | 8.8 (5.89) | 13.6 (6.65)
  Visit 5, n=123, 68, 116, 73 | 8.3 (7.12) [lower limit 7.12] | 12.6 (7.56) | 8.4 (5.89) | 12.8 (7.02)
  Visit 6, n=120, 66, 115, 74 | 7.4 (6.11) [lower limit 6.11] | 13.3 (8.26) | 8.5 (5.75) | 12.0 (7.52)
  Visit 7, n=120, 66, 113, 71 | 7.7 (6.51) [lower limit 6.51] | 12.4 (7.69) | 8.3 (6.48) | 11.4 (7.09)
  Visit 8, n=117, 66, 113, 70 | 7.2 (6.42) [lower limit 6.42] | 12.3 (7.56) | 7.8 (5.79) | 11.6 (7.70)

13. Secondary Outcome: Change From Baseline in CAT Total Score
Description: Participants were assessed for COPD symptoms by means of CAT at each Visit. This assessment was performed prior to the spirometry testing. A CAT total score of less than 10 represents best health status and greater than 15 represents worst health status. Baseline was the value at Visit 2 (randomization). Change from Baseline was calculated as specific timepoint value minus Visit 2 value. Scores were assessed at Visit 2 (Baseline), Visit 3 (Week 4), Visit 4 (Week 8), Visit 5 (Week 8), Visit 6 (Week 12), Visit 7 (Week 16), and Visit 8 (Week 24). Scores range from 0 to 40, high value in score indicate worse outcome.
Time Frame: Baseline and up to 24 weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SAL/FLU 50/250 µg BID-Single | SAL/FLU 50/250 µg BID-TRIPLE | TIO 18 µg QD-Single | TIO 18 µg QD-TRIPLE
Number analyzed (Participants) | 136 | 68 | 126 | 75
Scores on a scale
  Visit 3, n=132, 68, 121, 75 | -1.6 (4.74) | 0.1 (4.52) | 0.1 (3.97) | 2.1 (5.10)
  Visit 4, n=127, 68, 116, 74 | -1.7 (5.34) | -0.2 (5.68) | -0.3 (4.21) | 1.6 (5.53)
  Visit 5, n=123, 68, 116, 73 | -1.6 (6.04) | -0.8 (5.68) | -0.7 (5.14) | 0.8 (5.78)
  Visit 6, n=120, 66, 115, 74 | -2.3 (5.41) | 0.0 (6.28) | -0.7 (4.55) | 0.0 (6.09)
  Visit 7, n=120, 66, 113, 71 | -2.0 (5.50) | -0.8 (6.20) | -0.8 (4.91) | -0.6 (5.49)
  Visit 8, n=117, 66, 113, 70 | -2.4 (5.74) | -1.0 (6.05) | -1.4 (4.93) | -0.5 (6.29)

14. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1)
Description: FEV1 is defined as the volume of air forcefully expelled from the lungs in one second. At Screening (Visit 1) spirometric assessments were conducted before (Visit 1A) and 30 to 60 minutes after a bronchodilator challenge (400 µg of salbutamol) (Visit 1B). FEV1 during each visit are presented. FEV1 was assessed at Visit 1A (Screening), Visit 1B (Screening), Visit 2 (Baseline), Visit 3 (Week 4), Visit 4 (Week 8), Visit 5 (Week 8), Visit 6 (Week 12), Visit 7 (Week 16), and Visit 8 (Week 24).
Time Frame: Up to 24 weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | SAL/FLU 50/250 µg BID-Single | SAL/FLU 50/250 µg BID-TRIPLE | TIO 18 µg QD-Single | TIO 18 µg QD-TRIPLE
Number analyzed (Participants) | 136 | 68 | 126 | 75
Liters
  Visit 1A; n=136, 68, 126, 75 | 1.687 (0.4440) | 1.401 (0.4482) | 1.675 (0.4564) | 1.349 (0.4032)
  Visit 1B; n=136, 68, 126, 75 | 1.764 (0.4363) | 1.471 (0.4394) | 1.754 (0.4691) | 1.429 (0.4346)
  Visit 2; n=136, 68, 126, 75 | 1.695 (0.4650) | 1.385 (0.4336) | 1.681 (0.4929) | 1.362 (0.4267)
  Visit 3; n=131, 68, 119, 75 | 1.731 (0.4904) | 1.342 (0.4563) | 1.710 (0.5458) | 1.285 (0.4570)
  Visit 4; n=127, 68, 116, 74 | 1.713 (0.4943) | 1.355 (0.4555) | 1.703 (0.5215) | 1.336 (0.4638)
  Visit 5; n=122, 68, 116, 72 | 1.718 (0.4859) | 1.384 (0.4497) | 1.708 (0.5408) | 1.376 (0.4536)
  Visit 6; n=120, 66, 114, 74 | 1.716 (0.4817) | 1.413 (0.5104) | 1.712 (0.5353) | 1.405 (0.4938)
  Visit 7; n=119, 66, 113, 71 | 1.710 (0.4850) | 1.404 (0.4913) | 1.694 (0.5402) | 1.423 (0.4916)
  Visit 8; n=117, 66, 113, 70 | 1.694 (0.4808) | 1.435 (0.4871) | 1.688 (0.5426) | 1.390 (0.4695)

15. Secondary Outcome: Change From Baseline in FEV1
Description: FEV1 is defined as the volume of air forcefully expelled from the lungs in one second. Baseline was a value at Visit 2 (randomization). Change from Baseline was calculated as specific timepoint value minus Visit 2 value. FEV1 was assessed at Visit 2 (Baseline), Visit 3 (Week 4), Visit 4 (Week 8), Visit 5 (Week 8), Visit 6 (Week 12), Visit 7 (Week 16), and Visit 8 (Week 24).
Time Frame: Baseline (Visit 2) and up to 24 weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | SAL/FLU 50/250 µg BID-Single | SAL/FLU 50/250 µg BID-TRIPLE | TIO 18 µg QD-Single | TIO 18 µg QD-TRIPLE
Number analyzed (Participants) | 136 | 68 | 126 | 75
Liters
  Visit 3; n=131, 68, 119, 75 | 0.024 (0.1917) | -0.043 (0.1825) | 0.007 (0.1772) | -0.077 (0.1843)
  Visit 4; n=127, 68, 116, 74 | 0.008 (0.2092) | -0.030 (0.1821) | -0.011 (0.1977) | -0.032 (0.2325)
  Visit 5; n=122, 68, 116, 72 | -0.010 (0.2066) | -0.001 (0.1910) | -0.006 (0.2002) | 0.005 (0.2171)
  Visit 6; n=120, 66, 114, 74 | -0.007 (0.2069) | 0.027 (0.2025) | 0.002 (0.1893) | 0.037 (0.2098)
  Visit 7; n=119, 66, 113, 71 | -0.012 (0.2252) | 0.018 (0.1874) | -0.010 (0.2220) | 0.050 (0.2091)
  Visit 8; n=117, 66, 113, 70 | -0.019 (0.2293) | 0.049 (0.1892) | -0.017 (0.2355) | 0.027 (0.1999)

16. Secondary Outcome: Percentage of Participants Who Used Relief Medication (Salbutamol)
Description: Each evening participants recorded the number of occasions in the last 24 hours when they used their salbutamol for symptomatic relief of COPD symptoms. The percentage of participants who used relief medication in the study are presented.
Time Frame: 24 weeks
Population: mITT population
Measure: Number; unit: Percentage of participants
Arm/Group | SAL/FLU 50/250 µg BID-Single | SAL/FLU 50/250 µg BID-TRIPLE | TIO 18 µg QD-Single | TIO 18 µg QD-TRIPLE
Number analyzed (Participants) | 136 | 68 | 126 | 75
Percentage of participants | 40.4 | 61.8 | 43.7 | 70.7

17. Secondary Outcome: Percentage of Participants Who Stepped Down From TRIPLE Therapy to Initial Randomized Treatment
Description: The percentage of participants who stepped down from TRIPLE therapy to initial randomized treatment was calculated as number of participants who step-down from TRIPLE therapy divided by number of participants who switch to TRIPLE therapy and then multiplied by 100.
Time Frame: 24 weeks
Population: mITT population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TIO 18 µg QD | SAL/FLU 50/250 µg BID
Number analyzed (Participants) | 201 | 204
Percentage of participants | 1.33 [0.03 to 7.21] | 2.94 [0.36 to 10.22]

18. Secondary Outcome: Percentage of Participants Who Required Additional Treatment to TRIPLE Therapy
Description: The percentage of participants who required additional treatment to TRIPLE therapy is defined as number of participants who took additional medicine or therapy in TRIPLE therapy divided by number of participants who switch to TRIPLE therapy multiplied by 100.
Time Frame: 24 weeks
Population: mITT population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TIO 18 µg QD | SAL/FLU 50/250 µg BID
Number analyzed (Participants) | 201 | 204
Percentage of participants | 77.33 [66.21 to 86.21] | 72.06 [59.85 to 82.27]

19. Secondary Outcome: Percentage of Participants Who Dropped Out
Description: The percentage of participants who were withdrawn from the study.
Time Frame: 24 weeks
Population: All Subjects population: all participants who were enrolled into the study and whose data obtained at screening (visit1) was not missing and demography data was available.
Measure: Number; unit: Percentage of participants
Arm/Group | TIO 18 µg QD | SAL/FLU 50/250 µg BID
Number analyzed (Participants) | 202 | 204
Percentage of participants | 9 | 10

20. Secondary Outcome: Number of Participants in Each Treatment Efficacy Grade Evaluated by Participants
Description: Participants evaluated treatment efficacy by using the following grades: significantly improved (SII), moderately improved (MOI), mildly improved (MII), no change (NC), mildly worse (MIW), moderately worse (MOW), and significantly worse (SIW). Treatment efficacy was assessed at Visit 3 (Week 4), Visit 4 (Week 8), Visit 5 (Week 8), Visit 6 (Week 12), Visit 7 (Week 16), and Visit 8 (Week 24).
Time Frame: Up to 24 weeks
Population: mITT population
Measure: Number; unit: Participants
Arm/Group | SAL/FLU 50/250 µg BID-Single | SAL/FLU 50/250 µg BID-TRIPLE | TIO 18 µg QD-Single | TIO 18 µg QD-TRIPLE
Number analyzed (Participants) | 136 | 68 | 126 | 75
Participants
  Visit 3; SII | 5 | 0 | 1 | 1
  Visit 3; MOI | 9 | 2 | 3 | 3
  Visit 3; MII | 35 | 10 | 20 | 7
  Visit 3; NC | 74 | 32 | 85 | 32
  Visit 3; MIW | 7 | 19 | 9 | 22
  Visit 3; MOW | 1 | 5 | 3 | 9
  Visit 3; SIW | 1 | 0 | 0 | 1
  Visit 4; SII | 3 | 1 | 2 | 1
  Visit 4; MOI | 15 | 6 | 5 | 6
  Visit 4; MII | 31 | 12 | 25 | 21
  Visit 4; NC | 67 | 39 | 79 | 28
  Visit 4; MIW | 10 | 8 | 5 | 13
  Visit 4; MOW | 1 | 2 | 0 | 5
  Visit 5; SII | 2 | 1 | 2 | 4
  Visit 5; MOI | 13 | 7 | 3 | 6
  Visit 5; MII | 31 | 17 | 31 | 20
  Visit 5; NC | 66 | 34 | 78 | 31
  Visit 5; MIW | 10 | 7 | 2 | 9
  Visit 5; MOW | 0 | 2 | 0 | 3
  Visit 5; SIW | 1 | 0 | 0 | 0
  Visit 6; SII | 2 | 1 | 2 | 4
  Visit 6; MOI | 13 | 4 | 4 | 13
  Visit 6; MII | 35 | 16 | 30 | 14
  Visit 6; NC | 66 | 33 | 72 | 34
  Visit 6; MIW | 4 | 11 | 7 | 7
  Visit 6; MOW | 0 | 0 | 0 | 2
  Visit 6; SIW | 0 | 1 | 0 | 0
  Visit 7; SII | 1 | 2 | 2 | 4
  Visit 7; MOI | 13 | 4 | 5 | 11
  Visit 7; MII | 27 | 17 | 28 | 20
  Visit 7; NC | 75 | 37 | 71 | 26
  Visit 7; MIW | 4 | 5 | 7 | 9
  Visit 7; MOW | 0 | 1 | 0 | 1
  Visit 8; SII | 5 | 1 | 2 | 4
  Visit 8; MOI | 9 | 4 | 8 | 9
  Visit 8; MII | 39 | 19 | 30 | 19
  Visit 8; NC | 58 | 37 | 69 | 34
  Visit 8; MIW | 5 | 5 | 3 | 4
  Visit 8; MOW | 1 | 0 | 1 | 0

21. Secondary Outcome: Number of Participants in Each Treatment Efficacy Grade Evaluated by Physician
Description: Physician evaluated treatment efficacy by using the following grades: significantly improved (SII), moderately improved (MOI), mildly improved (MII), no change (NC), mildly worse (MIW), moderately worse (MOW), and significantly worse (SIW). Treatment efficacy was assessed at Visit 3 (Week 4), Visit 4 (Week 8), Visit 5 (Week 8), Visit 6 (Week 12), Visit 7 (Week 16), and Visit 8 (Week 24).
Time Frame: 24 weeks
Population: mITT population
Measure: Number; unit: Participants
Arm/Group | SAL/FLU 50/250 µg BID-Single | SAL/FLU 50/250 µg BID-TRIPLE | TIO 18 µg QD-Single | TIO 18 µg QD-TRIPLE
Number analyzed (Participants) | 136 | 68 | 126 | 75
Participants
  Visit 3; SII | 6 | 0 | 1 | 1
  Visit 3; MOI | 11 | 1 | 5 | 4
  Visit 3; MII | 40 | 12 | 21 | 3
  Visit 3; NC | 67 | 31 | 83 | 32
  Visit 3; MIW | 7 | 16 | 7 | 23
  Visit 3; MOW | 0 | 8 | 3 | 12
  Visit 3; SIW | 1 | 0 | 1 | 0
  Visit 4; SII | 3 | 1 | 2 | 0
  Visit 4; MOI | 14 | 3 | 8 | 9
  Visit 4; MII | 28 | 13 | 23 | 18
  Visit 4; NC | 74 | 33 | 79 | 27
  Visit 4; MIW | 6 | 12 | 4 | 12
  Visit 4; MOW | 1 | 6 | 0 | 8
  Visit 4; SIW | 1 | 0 | 0 | 0
  Visit 5; SII | 1 | 2 | 2 | 4
  Visit 5; MOI | 12 | 6 | 4 | 8
  Visit 5; MII | 29 | 14 | 22 | 19
  Visit 5; NC | 73 | 35 | 83 | 29
  Visit 5; MIW | 7 | 10 | 5 | 10
  Visit 5; MOW | 0 | 1 | 0 | 3
  Visit 5; SIW | 1 | 0 | 0 | 0
  Visit 6; SII | 2 | 1 | 2 | 2
  Visit 6; MOI | 10 | 1 | 3 | 11
  Visit 6; MII | 31 | 18 | 28 | 17
  Visit 6; NC | 74 | 33 | 72 | 32
  Visit 6; MIW | 3 | 11 | 10 | 9
  Visit 6; MOW | 0 | 1 | 0 | 3
  Visit 6; SIW | 0 | 1 | 0 | 0
  Visit 7; SII | 0 | 1 | 2 | 3
  Visit 7; MOI | 13 | 2 | 5 | 12
  Visit 7; MII | 25 | 18 | 23 | 12
  Visit 7; NC | 79 | 38 | 77 | 35
  Visit 7; MIW | 3 | 5 | 5 | 8
  Visit 7; MOW | 0 | 2 | 1 | 1
  Visit 8; SII | 2 | 1 | 3 | 3
  Visit 8; MOI | 7 | 4 | 7 | 9
  Visit 8; MII | 36 | 19 | 27 | 13
  Visit 8; NC | 70 | 39 | 71 | 40
  Visit 8; MIW | 1 | 2 | 4 | 5
  Visit 8; MOW | 1 | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events and non-serious adverse events were collected from the start of study treatment and until the follow up contact (up to Week 26).
Description: Serious adverse events and non-serious adverse events were reported for Safety population
Arm/Group | TIO 18 µg QD-Single | TIO 18 µg QD-TRIPLE | SAL/FLU 50/250 µg BID-Single | SAL/FLU 50/250 µg BID-TRIPLE
Serious Adverse Events (participants affected / at risk) | 8/126 | 8/75 | 8/136 | 6/68
Other Adverse Events (participants affected / at risk) | 29/126 | 29/75 | 48/136 | 25/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TIO 18 µg QD-Single (N=126) | TIO 18 µg QD-TRIPLE (N=75) | SAL/FLU 50/250 µg BID-Single (N=136) | SAL/FLU 50/250 µg BID-TRIPLE (N=68)
Pneumonia (Infections and infestations) | 0 | 2 | 2 | 2
Bronchopneumonia (Infections and infestations) | 0 | 1 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Liver abscess (Infections and infestations) | 0 | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Anal polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 0
Varicose vein (Vascular disorders) | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Disuse syndrome (General disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TIO 18 µg QD-Single (N=126) | TIO 18 µg QD-TRIPLE (N=75) | SAL/FLU 50/250 µg BID-Single (N=136) | SAL/FLU 50/250 µg BID-TRIPLE (N=68)
Nasopharyngitis (Infections and infestations) | 19 | 20 | 25 | 14
Bronchitis (Infections and infestations) | 6 | 5 | 7 | 7
Pneumonia (Infections and infestations) | 0 | 4 | 2 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 18 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.